CLINICAL TRIAL: NCT03531593
Title: Dose Effect Relationship of Methotrexate and Hepatic Fibrosis in Patients With Inflammatory Bowel Disease
Brief Title: Dose Effect Relationship of MTX and IBD
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: 16040304
Record Dates: First submitted 2017-04-26; First posted 2018-05-22 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Inflammatory Bowel Diseases; Liver Fibroses; Methotrexate
Keywords: MTX; IBD; US Elastography; Liver Fibrosis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- US Elastography: All subjects will undergo one ultrasound elastography examination after consent.
  Interventions: Diagnostic Test: Ultrasound Elastography

INTERVENTIONS:
Diagnostic Test: Ultrasound Elastography — Ultrasound elastography is a new, noninvasive technique that can assess the stiffness of the liver by the evaluation of how sound waves propagate through the liver parenchyma.

SUMMARY:
Currently there are no guidelines for monitoring hepatic fibrosis associated with long term MTX use. Routine liver biopsies are not being done as a part of surveillance due to potential complications like bleeding and pneumothorax. Non-invasive markers like gammaglamyltransferase (GGTP), Alkaline Phosphatase (AlkPhos), Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are deranged at a late stage and may not be helpful in detecting early fibrosis. The current study will utilize a sensitive, but noninvasive, test to evaluate for hepatic fibrosis. We are attempting to screen for early detection of fibrosis due to MTX before it progresses to irreversible cirrhosis and end-stage liver disease. Based on the results of this pilot study, ultrasound elastography could be used to prospectively study a larger population to establish guidelines for monitoring safety and hepatic complications with MTX. The influence of other co-morbid factors like obesity, alcohol ingestion and smoking is critical to identifying high risk patients who may require closer monitoring. We follow close to 550 patients with IBD. If we presume that at least 20% patients are currently receiving methotrexate, we will be able to recruit enough patients for this pilot study.

DETAILED DESCRIPTION:
Inflammatory bowel disease is a chronic, relapsing and remitting, inflammatory disorder of the GI tract. The mainstay of medical therapy is comprised of 5-aminosalicylates, corticosteroids, immunomodulators such as mercaptopurine and MTX, and biologics such as infliximab and adalimumab.

Mercaptopurine historically had been the immunomodulator of choice for disease maintenance and as an adjuvant to biologic therapy to prevent antibody formation.

However in 2008 the FDA communicated an increase incidence of a lethal blood cancer, hepatosplenic T-cell lymphoma, in adolescent males taking mercaptopurine along with Infliximab. In addition there is a known four-fold increase in the risk of lymphoma in patients treated with mercaptopurine while the risk is not significantly increased with MTX use. Due to these reasons there has been a shift amongst pediatric gastroenterologists to starting children with newly diagnosed IBD on MTX as a first line immunomodulator and/or as an adjuvant to biologic therapy. Given the chronic nature of this disease, children are more likely to be on long term MTX therapy. There is paucity of data for evaluation and monitoring of hepatic fibrosis associated with prolonged methotrexate usage in patients with IBD. The influence of co-morbid factors like obesity, alcohol intake and smoking are also not well understood. The primary purpose of this pilot study is to assess for hepatic fibrosis using shear wave elastography in patients on methotrexate in relation to the cumulative dose they have received. .

MTX is a folic acid antagonist, which has been used as a mainstay of therapy in other chronic inflammatory diseases such as rheumatoid arthritis and psoriatic arthritis. Known side effects from the medication are nausea, leukopenia and hepatotoxicity. In addition, patients with refractory psoriasis on MTX therapy are reported to develop hepatic fibrosis in a cumulative dose dependent fashion. Currently the gold standard of assessment is a liver biopsy, as serological biomarkers have proven to correlate poorly in early stages of fibrosis. Liver biopsy is not only an invasive test but could lead to serious complications such as pneumothorax and intra-peritoneal bleeding.

As standard of care our pediatric patients with IBD on MTX therapy are screened quarterly with serological biomarkers such as complete blood counts, albumin and liver function tests to evaluate for these side effects. As previously stated, the dilemma arises in that the derangement of these lab tests poorly correlate with early stages of fibrosis and it is likely that by the time they are elevated the patient already has experienced irreversible liver damage. In fact in an adult study by Te et al in 2000 reported that patients with IBD on MTX show poor correlation of liver function tests and histological findings on liver biopsy. Therefore they concluded that following the same surveillance guidelines in IBD patients on MTX as those with psoriasis on MTX is not warranted as risks of the procedure outweigh the benefits of biopsy. Pediatric patients with a lifelong diagnosis of IBD and a life expectancy of 80 years can reach a considerably higher cumulative MTX dose over their lifetime and may need non-invasive monitoring for liver damage and fibrosis.

Ultrasound elastography is a new, noninvasive technique that can assess the stiffness of the liver by the evaluation of how sound waves propagate through the liver parenchyma. It can evaluate multiple areas of the liver in contrast to liver biopsy that only can sample a small area of tissue. Sampling of multiple areas of the liver is helpful in heterogeneous distribution of liver disease. Several recent studies have demonstrated the superiority of shear wave elastography over other older ultrasound based methods. A recent study also demonstrated reliability of detecting hepatic fibrosis in children using shearwave elastography and correlating with simultaneously obtained liver biopsies (7) Shear wave ultrasound elastography is a quantitative subset of ultrasound elastography that has good reproducibility and has good sensitivity/specificity for assessing for severe fibrosis and cirrhosis. A recent report by Tae Yeob Kim et al (demonstrated hepatic fibrosis in 5% patients on long term methotrexate for rheumatoid arthritis which was associated with high body mass index rather than cumulative methotrexate dose).(8) There are no similar studies in children or adults with IBD.

2. RATIONALE Currently there are no guidelines for monitoring hepatic fibrosis associated with long term MTX use. Routine liver biopsies are not being done as a part of surveillance due to potential complications like bleeding and pneumothorax. Non-invasive markers like gammaglamyltransferase (GGTP), Alkaline Phosphatase (AlkPhos), Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are deranged at a late stage and may not be helpful in detecting early fibrosis. The current study will utilize a sensitive, but noninvasive, test to evaluate for hepatic fibrosis. We are attempting to screen for early detection of fibrosis due to MTX before it progresses to irreversible cirrhosis and end-stage liver disease. Based on the results of this pilot study, ultrasound elastography could be used to prospectively study a larger population to establish guidelines for monitoring safety and hepatic complications with MTX. The influence of other co-morbid factors like obesity, alcohol ingestion and smoking is critical to identifying high risk patients who may require closer monitoring. We follow close to 550 patients with IBD. If we presume that at least 20% patients are currently receiving methotrexate, we will be able to recruit enough patients for this pilot study.

STUDY DESIGN

This is a single site prospective cross-sectional pilot study that will aim to enroll IBD patients who have different cumulative dose exposures to MTX. Each patient who consents will undergo an ultrasound elastography exam. We will aim to enroll an equal number of patients in four categories (25 each) based on lifetime cumulative MTX dose:

Category Lifetime cumulative MTX dose (g) 0 (Control Group) No MTX, but DX of IBD

1. 0-1.5
2. 1.5-3
3. >3

3. TARGET STUDY POPULATION SPECIFICS Inclusion Criteria

• Patients age 2-22 years of age who have a diagnosis of IBD and consent to our study.

Exclusion Criteria

* Patient is unable to tolerate an ultrasound elastography examination.
* Target enrollment for the MTX dose category in which the patient fits has been completed.
* Any preexisting liver disease

  4. DATA COLLECTION Data Collection Procedures Candidates for the study will be identified by the Gastroenterology service or self-refer in response to advertisements and will be consented by one of the members of the research team. Consented subjects will be scheduled for research ultrasound elastography examination at CMH. Dr. Chan, Pediatric Radiologist and Co-Investigator, will review the ultrasound elastography images for shear wave velocity. Demographic and clinical variables will be collected from the chart at the time of enrollment and ultrasound elastography examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 2-22 years of age who have a diagnosis of IBD and consent to our study.

Exclusion Criteria:

* Patient is unable to tolerate an ultrasound elastography examination.
* Target enrollment for the MTX dose category in which the patient fits has been completed.
* Any preexisting liver disease

Ages: 2 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients ages 2-22 whom have a diagnosis of IBD can participate in our study. We will recruit a total of 100 subjects; 25 control subjects and 75 subjects whom are taking Methotrexate for their IBD.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Primary Objective - correlation between velocities of shear wave elastography and cumulative dose of Methotrexate (MTX) in patients with Inflammatory Bowel Disease (IBD). | 2/1/2017-10/31/2017
  To evaluate the correlation between velocities of shear wave elastography and cumulative dose of Methotrexate (MTX) in patients with Inflammatory Bowel Disease (IBD).

SECONDARY OUTCOMES:
Secondary Objective - correlate hepatic enzymes elevation and ultrasound elastography velocities | 2/1/2017-10/31/2017
  To correlate hepatic enzymes elevation and ultrasound elastography velocities.
Third Objective - changes in shear wave velocity | 2/1/2017-10/31/2017
  To assess if changes in shear wave velocity due to Methotrexate are influenced by other risk factors like obesity, alcohol ingestion, smoking
Fourth Objective - correlate ultrasound elastography findings with fibrosis markers | 2/1/2017-10/31/2017
  To correlate ultrasound elastography findings with fibrosis markers: AST/ALT ratio (AST (U/L0/ALT (U/L); AST/platelet ratio index (AST/upper limit of normal)/Platelet count (109/L) X 100

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Asrani SK. Incorporation of Noninvasive Measures of Liver Fibrosis Into Clinical Practice: Diagnosis and Prognosis. Clin Gastroenterol Hepatol. 2015 Nov;13(12):2190-204. doi: 10.1016/j.cgh.2015.07.030. Epub 2015 Jul 27. PMID 26226095
- [Result] Barbero-Villares A, Mendoza Jimenez-Ridruejo J, Taxonera C, Lopez-Sanroman A, Pajares R, Bermejo F, Perez-Calle JL, Mendoza JL, Algaba A, Moreno-Otero R, Mate J, Gisbert JP; Madrid Group for the Study of Inflammatory Bowel Disease ENICMAD. Evaluation of liver fibrosis by transient elastography (Fibroscan(R)) in patients with inflammatory bowel disease treated with methotrexate: a multicentric trial. Scand J Gastroenterol. 2012 May;47(5):575-9. doi: 10.3109/00365521.2011.647412. Epub 2012 Jan 10. PMID 22229701
- [Result] Bota S, Paternostro R, Etschmaier A, Schwarzer R, Salzl P, Mandorfer M, Kienbacher C, Ferlitsch M, Reiberger T, Trauner M, Peck-Radosavljevic M, Ferlitsch A. Performance of 2-D shear wave elastography in liver fibrosis assessment compared with serologic tests and transient elastography in clinical routine. Ultrasound Med Biol. 2015 Sep;41(9):2340-9. doi: 10.1016/j.ultrasmedbio.2015.04.013. Epub 2015 May 23. PMID 26004669
- [Result] Khan N, Abbas AM, Whang N, Balart LA, Bazzano LA, Kelly TN. Incidence of liver toxicity in inflammatory bowel disease patients treated with methotrexate: a meta-analysis of clinical trials. Inflamm Bowel Dis. 2012 Feb;18(2):359-67. doi: 10.1002/ibd.21820. Epub 2011 Jul 12. PMID 21751301
- [Result] Te HS, Schiano TD, Kuan SF, Hanauer SB, Conjeevaram HS, Baker AL. Hepatic effects of long-term methotrexate use in the treatment of inflammatory bowel disease. Am J Gastroenterol. 2000 Nov;95(11):3150-6. doi: 10.1111/j.1572-0241.2000.03287.x. PMID 11095334
- [Result] Valentino PL, Church PC, Shah PS, Beyene J, Griffiths AM, Feldman BM, Kamath BM. Hepatotoxicity caused by methotrexate therapy in children with inflammatory bowel disease: a systematic review and meta-analysis. Inflamm Bowel Dis. 2014 Jan;20(1):47-59. doi: 10.1097/01.MIB.0000436953.88522.3e. PMID 24280876
- [Result] Dillman JR, Heider A, Bilhartz JL, Smith EA, Keshavarzi N, Rubin JM, Lopez MJ. Ultrasound shear wave speed measurements correlate with liver fibrosis in children. Pediatr Radiol. 2015 Sep;45(10):1480-8. doi: 10.1007/s00247-015-3345-5. Epub 2015 Apr 8. PMID 25851300
- [Result] Kim TY, Kim JY, Sohn JH, Lee HS, Bang SY, Kim Y, Kim MY, Jeong WK. Assessment of Substantial Liver Fibrosis by Real-time Shear Wave Elastography in Methotrexate-Treated Patients With Rheumatoid Arthritis. J Ultrasound Med. 2015 Sep;34(9):1621-30. doi: 10.7863/ultra.15.14.10035. Epub 2015 Aug 12. PMID 26269292
- [Result] Malatjalian DA, Ross JB, Williams CN, Colwell SJ, Eastwood BJ. Methotrexate hepatotoxicity in psoriatics: report of 104 patients from Nova Scotia, with analysis of risks from obesity, diabetes and alcohol consumption during long term follow-up. Can J Gastroenterol. 1996 Oct;10(6):369-75. doi: 10.1155/1996/213596. PMID 9193771